CLINICAL TRIAL: NCT04667741
Title: A Comparative Study Between Turkey and Portugal: Post-dialysis Recovery Time and Affecting Factors
Brief Title: Post-dialysis Recovery Time and Affecting Factors Between Turkey and Portugal
Status: Completed | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Other Study IDs: 12869
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Dialysis; Recovery Time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Post-dialysis recovery group — Before the hemodialysis session, the patients were asked by the investigators how long it took them to recover from a dialysis session, taking the last treatment month into account.

SUMMARY:
Patients undergoing hemodialysis (HD) can experience symptoms such as lassitude, pain, muscle cramps, nausea, vomiting, constipation, diarrhea, rash, skin dryness, sleep disorders, and emotional and sexual problems after the treatment.

DETAILED DESCRIPTION:
Many chronic HD patients do not feel well after the treatment sessions and need some time to recover. This recovery time is defined as the time required to recover from the feelings of lassitude and fatigue. The patients are limited in their daily living activities at home and at work during this period and a significant amount of time is therefore required to go back to normal life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Being on HD for 4 hours a day on 3 days per week for at least 6 months
* No communication problem
* Volunteering to participate to the study

Exclusion Criteria:

* Younger than 18 years
* Shorter being on HD for 4 hours a day on 3 days per week for at least 6 months
* Have communication problem
* Not volunteering to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being on HD for 4 hours a day on 3 days per week for at least 6 months and 18 years or older in turkey and Portugal
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Post-dialysis Recovery Time | up to 4 weeks
  Before the hemodialysis session, the patients were asked by the investigators how long it took them to recover from a dialysis session, taking the last treatment month into account.
Anxiety at one month | up to 4 weeks
  It will be assessed with Hospital Anxiety and Depression Scale. This scale, which has a two-factor structure is comprised of 14 items. Seven of these items assess the anxiety status and the remaining seven assess depression.
  Each item is scored on a four-point scale. Total score ranges between 0 and 21 for anxiety and depression. Scores between 0 and 7 indicate normal emotional status.
Depression at one month | up to 4 weeks
  It will be assessed with Hospital Anxiety and Depression Scale. This scale, which has a two-factor structure is comprised of 14 items. Seven of these items assess the anxiety status and the remaining seven assess depression.
  Each item is scored on a four-point scale. Total score ranges between 0 and 21 for anxiety and depression. Scores between 0 and 7 indicate normal emotional status.
Rate of Headache at one month | up to 4 weeks
  The patients will tell the living of headache to the investigators at the end of the one month. The answer will be "yes" or "no".
Rate of dry mouth at one month | up to 4 weeks
  The patients will tell the living of dry mouth to the investigators at the end of the one month. The answer will be "yes" or "no".
Rate of trouble falling asleep at one month | up to 4 weeks
  The patients will tell the living of trouble falling asleep to the investigators at the end of the one month. The answer will be "yes" or "no".
Hemodialysis Sessions Features | up to 4 weeks
  Before and after the hemodialysis sessions, the patients were asked by investigators about dialysate bicarbonate concentration in mmol/L
Biochemical variables at one month | up to 4 weeks
  After one month urea reduction rate (%) were aken from the patients' medical record

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Assoc. Prof., Study Director — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umeukeje EM, Cavanaugh KL. Intradialytic Symptoms and Recovery Time: Thinking 'Outside the Box' to Improve Patients' Dialysis Experience. Kidney Med. 2020 Feb 28;2(2):98-101. doi: 10.1016/j.xkme.2020.02.001. eCollection 2020 Mar-Apr. No abstract available. PMID 32734955
- [Background] Alvarez L, Brown D, Hu D, Chertow GM, Vassalotti JA, Prichard S. Intradialytic Symptoms and Recovery Time in Patients on Thrice-Weekly In-Center Hemodialysis: A Cross-sectional Online Survey. Kidney Med. 2019 Dec 20;2(2):125-130. doi: 10.1016/j.xkme.2019.10.010. eCollection 2020 Mar-Apr. PMID 32734233
- [Background] Bossola M, Di Stasio E, Monteburini T, Parodi E, Ippoliti F, Cenerelli S, Santarelli S, Nebiolo PE, Sirolli V, Bonomini M, Antocicco M, Zuccala G, Laudisio A. Recovery Time after Hemodialysis Is Inversely Associated with the Ultrafiltration Rate. Blood Purif. 2019;47(1-3):45-51. doi: 10.1159/000492919. Epub 2018 Sep 19. PMID 30231240
- [Derived] Ozen N, Eyileten T, Teles P, Seloglu B, Gurel A, Ocuk A, Ozen V, Fernandes F, Campos L, Coutinho S, Teixeira J, Moura SCM, Ribeiro O, Sousa CN. Impact of variables on recovery time in patients undergoing hemodialysis: an international survey. BMC Nephrol. 2025 Jan 8;26(1):13. doi: 10.1186/s12882-024-03937-9. PMID 39780078